CLINICAL TRIAL: NCT07394283
Title: Impact of Night Shift Work on Dietary Habits Among Intensive Care and Emergency Healthcare Workers: An Observational Questionnaire-Based Study
Brief Title: Impact of Night Shift Work on Dietary Habits Among Intensive Care and Emergency Healthcare Workers (NUTRINIGHT)
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 26Onco-Hémato01
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Shift-work Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare Night Shift Workers
  Interventions: Other: Healthcare Night Shift Workers
- Non-Healthcare Night Shift Workers
  Interventions: Other: Healthcare Night Shift Workers

INTERVENTIONS:
Other: Healthcare Night Shift Workers — Data are collected through an anonymous, self-administered online questionnaire.

SUMMARY:
Night shift work is an essential component of healthcare systems, particularly in intensive care units and emergency departments, where continuous patient monitoring and rapid clinical decision-making are required. However, it is associated with diruption of the circadian rhythm , sleep disturbances, and physiological stress, which may influence lifestyle behaviors, including dietary habits. Previous studies have reported that night work can be associated with changes in meal timing, increased caloric intake, preference for energy-dense foods, and reduced overall diet quality.Despite the growing literature on night work and nutrition, data specifically describing dietary habits among healthcare professionals working night shifts in high-intensity clinical settings remain limited. Intensive care units and emergency departments combine high workload, psychological stress, time constraints, and restricted access to appropriate meals during night hours, all of which may affect eating behaviors. Moreover, whether these dietary patterns are specific to healthcare professionals or primarily related to night work itself remains unclear. This observational, cross-sectional study aims to describe dietary habits among healthcare professionals working night shifts in intensive care units and emergency departments, and to compare these habits with those of night workers from non-healthcare sectors. Data will be collected prospectively through a voluntary, anonymous, self-administered online questionnaire during a defined inclusion period. The questionnaire will explore meal timing, eating patterns, food choices, and constraints perceived as influencing dietary behaviors during night work. By providing a descriptive overview of dietary habits across different categories of night workers, the study seeks to improve understanding of how night work and occupational context influence eating behaviors. The findings may contribute to the development of future preventive strategies and workplace health initiatives aimed at improving the health and well-being of night shift workers

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Currently working night shifts.
* Employment in healthcare (intensive care units or emergency departments) or in non-healthcare professional sectors
* Voluntary participation and completion of the online questionnaire

Exclusion Criteria:

* None

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of adult night shift workers from different professional sectors. This includes healthcare professionals working in intensive care units and emergency departments, as well as night workers employed innon-healthcare sectors. Participation is voluntary, and data are collected through an anonymous, self-administered online questionnaire."
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Dietary Habits of Night Shift Workers | At the inclusion
  Online questionnaire without score

SECONDARY OUTCOMES:
Meal Timing During Night Shifts | At the inclusion
  Anonymous self-administered online questionnaire without score
Eating Patterns During Night Shifts | At the inclusion
  Anonymous self-administered online questionnaire without score
Comparison of Dietary Habits Between Healthcare and Non-Healthcare Night Shift Workers | At the inclusion
  Questionnaire data

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Alpes-Maritimes, France